CLINICAL TRIAL: NCT07360236
Title: Determining the Effect of Shoulder Flexion Angle on Latissimus Dorsi and Forearm Flexor Hypertrophy
Acronym: LPDLR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Cameron Mitchell, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H25-03685
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Muscle Hypertrophy; Muscular Strength
Keywords: Muscle hypertrophy; Long muscle length; Short muscle length; Range of motion; Muscular strength; 1RM; Length-tension Relationship; Resistance Training; Neuromechanical Matching; Latissimus dorsi; Lat Pulldown; Lat Row

STUDY DESIGN:
Intervention Model Description: Within-Subject Design: Each participant will have the left and right arm randomly assigned to the either LAT PULLDOWN or LAT ROW condition. Each participant will perform both conditions, exclusively for the left or right arm. This helps to control for genetics, nutrition, recovery, stress management and training history as each participant acts as a self-control group as well as both experimental conditions.
Masking Description: The MRi analyst will be blinded to the the unique participant code assigned to each MRi file when measuring cross sectional area and muscle volume. Another member of the research group will assign random numbers to each copy of the MRi files that are measured by the MRi analyst.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LAT PULLDOWN and LAT ROW Training Protocol (Experimental): Using a within subject design, participants will have the arms from both left and right side of the body (divided by sagittal plane) randomly assigned to either LAT PULLDOWN or LAT ROW conditions. Participants will then engage in maximal strength testing on the Lat Pulldown and Lat Row cable machines (1RM) as well as isokinetic strength testing (1080 Quantum Syncro) in weeks 1 and 12. Participants will engage in the LAT PULLDOWN and LAT ROW training sessions for 10 weeks in duration from week 2 until week 11.
  Interventions: Other: LAT PULLDOWN and LAT ROW training sessions; Other: Maximal isotonic strength testing (1RM); Other: Isokinetic strength testing (1080 Quantum)

INTERVENTIONS:
Other: LAT PULLDOWN and LAT ROW training sessions — One arm will be randomly assigned to perform LAT PULLDOWN and the contralateral arm will be randomly assigned to perform LAT ROW on a cable machine. Each exercise will include 1 warm up set at 50% 1RM followed by 4-5 sets of 8-12 repetitions per limb. 2 minutes of rest between sets on the ipsilateral limb with 30s between the contralateral limb. The left and right limbs will alternate each session in which one starts each exercise, resulting in 10 training sessions each where the left and right limbs starts first on each exercise. All sets will be performed to momentary failure. A Dynamic Double Progression will be employed to ensure intensity is maintained throughout the intervention.
Other: Maximal isotonic strength testing (1RM) — Each limb will perform a 1RM strength test of the Lat Pulldown and Lat Row on the cable machine respectively. Testing will occur in weeks 1 and 12 of the study with the non-dominant arm tested before the dominant arm. Participants self-selects first warm up set with a weight that is performed between 6-10 repetitions on both limbs. Rest for 1 minute between limbs and subsequent set. A weight is then selected by research staff to perform 3 repetitions with based on previous set. Load is now increased until 1RM is achieved. 3 minutes of rest will be taken between 1RM attempts, with 1RM being complete within 3-5 attempts. Participant will rest 3 minutes before starting testing on the other exercise. The 1RM protocol is repeated for the second exercise. Initial strength testing results and progression from the 10 week training intervention will help to inform testing weights for the post strength testing session. Post strength testing will follow the same protocol as pre strength testing.
Other: Isokinetic strength testing (1080 Quantum) — Participants will engage in isokinetic strength testing on the 1080 Quantum Syncro machine in weeks 1 and 12 for both movements: Shoulder extension from 180° and shoulder extension from 90°. Participants will perform each movement unilaterally. Participants will start with the non-dominant arm. Each movement will be tested through A maximal active range of motion. Participants will complete 10 sub-maximal repetitions to allow familiarization each movement. After a 2-minute rest, participants will complete 4 maximal concentric and eccentric repetitions with 3 minutes rest at 30°/second for 3 sets. The protocol is then repeated on the dominant limb.

SUMMARY:
The goal of this clinical trial is to learn the effect of training a muscle at a longer or shorter muscle length during resistance exercise in young and healthy adults. Participants will undergo two types of resistance training conditions that are randomly assigned to the left and right arm. The LATPULLDOWN (LPD) condition refers to performing an exercise that places the latissimus dorsi muscle at a long muscle length when the shoulder is elevated to 180° of shoulder flexion. The LATROW (LR) condition refers to performing an exercise that places the latissimus dorsi muscle at a shorter muscle length when the shoulder is elevated to 90° of shoulder flexion.

The main questions the trial aims to answer are:

1. Does resistance training the latissimus dorsi muscle at a long muscle length result in greater muscle growth than training at a shorter muscle length?
2. Does resistance training the latissmus dorsi muscle at long or short muscle lengths result in regional muscle growth differences of the latissimus dorsi?

We hypothesize that:

1. LAT PULLDOWN will induce greater hypertrophy compared to LAT ROW condition
2. LAT PULLDOWN will result in greater increases in 1RM compared to LATROW condition
3. LAT PULLDOWN and LAT ROW will result in angle specific differences in Isokinetic strength
4. LAT PULLDOWN will result in greater inferior Latissimus Dorsi hypertrophy
5. LAT ROW will result in greater superior Latissimus Dorsi hypertrophy

The investigators will compare the change in muscle volume and muscular strength between the LAT PULLDOWN and LAT ROW training conditions, which each participant will have the left and right arm randomly assigned to either exclusively LAT PULLDOWN or LAT ROW conditions.

Participants will:

* Resistance train the left and right arm with two separate conditions; LAT PULLDOWN and LAT ROW for 12 weeks, with the first and last weeks dedicated to only strength testing (Isotonic and Isokinetic) and measuring muscle volume via magnetic resonance imaging (MRI)
* Visit the gym for resistance training 2 times per week
* Visit the UBC MRI Research Facility in weeks 1 and 12 for MRI of muscle volume

DETAILED DESCRIPTION:
Statistical Analysis:

Null Hypothesis Significance Testing (NHST) will be used to measure differences in hypertrophy, differences in 1RM strength and isokinetic strength between LAT PULLDOWN and LAT ROW conditions.

It is anticipated that this study will require at least 20 participants to be screened and registered into the trial. Data will be analyzed on the basis that all participants will be included in the analysis. Participants who drop out (withdraw from treatment) will be followed up with to collect all available data and will not be replaced. Missing data will be assumed missing at random.

Sample Size Calculation:

Based on the effect size reported by Maeo et al. (2023) for difference in triceps brachia long head hypertrophy between training performed in the lengthened compared to shortened position using a within participant design, (d=0.61) a sample size of 20 participants was calculated to achieve an a priori power of 90%.

ELIGIBILITY:
Inclusion Criteria:

1. Any sex
2. Able to understand and communicate in English
3. 19-30 years of age
4. All "No" answers on the CSEP Get Active questionnaire or doctors' approval to participate
5. Trained participants: Structured resistance training over at least the past 12-months (i.e., ≥ 2 hours per week of structured/periodized training)

Exclusion Criteria:

Participants will be excluded from this study if they meet any of the following criteria:

1. BMI lower than 18 or greater than 30
2. Difficulty to understand and communicate in English
3. Current use of cigarettes or other nicotine devices
4. Any major uncontrolled cardiovascular, muscular, metabolic, and/or neurological disorders
5. Any medical condition impacting the ability to participate in maximal exercise
6. Type one or type two diabetes
7. Diagnosis of cancer or undergoing cancer treatment in the past 12 months
8. Drug therapy with any drugs that alter skeletal muscle metabolism (i.e., Metformin, Benzodiazepines)
9. Implants containing ferrous metal
10. Surgery or tattoos (including tattooed eyeliner) in the last 6 weeks
11. Pregnancy

Magnetic Resonance Imaging (MRI) Exclusion Criteria

CANNOT participate if you have any of the following:

1. Retained wires from an electronic implant that has been removed (i.e., pacemaker wires not attached to a pacemaker)
2. Cardiac pacemaker or defibrillator
3. Metal in eye or orbit
4. Ferromagnetic aneurysm clip
5. Makeup tattoos that are not designed to fade over time
6. Stainless steel intrauterine device (IUD)

Depending on the individual situation, you may not be able to participate if you have/had any of the following:

1. Artificial heart valve
2. Ear or eye implant
3. Brain aneurysm clip
4. Implanted electronic device (i.e., drug infusion pump, electrical stimulator)
5. Orthopedic hardware (artificial joint, plate, screw, rod)
6. Shrapnel, bullets, or other metal fragments
7. Surgery, medical procedure, or tattoos (including tattooed eyeliner) in the last six weeks
8. Other metallic prostheses

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Muscle volume and Cross sectional area | From enrolment to the end of the intervention at 12 weeks
  Muscle volume of the latissimus dorsi, biceps brachii, brachialis, posterior deltoid and teres major muscle will be measured by cross sectional area (CSA) via Magnetic Resonance Imaging (MRI). The entire muscle length will be imaged and images at 25%, 50% and 75% of the entire muscle length will be analyzed to calculate CSA and any regional differences in hypertrophy.

SECONDARY OUTCOMES:
Isotonic strength testing (1RM) | Initial testing in week 1 and final testing in week 12
  Isotonic strength testing will compare the magnitude of gains in isotonic strength via a one repetition maximum test (1RM) which is the maximum weight lifted for 1 repetition. Isotonic strength will be measured using a cable machine for a Lat Pulldown and Lat Row exercise. Single arm shoulder extension from 180° and 90° will be tested for 1RM (maximum weight lifted for 1 repetition).
Isokinetic strength testing | Initial testing in week 1 to final testing in week 12
  Isokinetic Strength Testing: Compare the magnitude of gains in isokinetic strength in the LAT PULLDOWN and LAT ROW conditions for two movements. Single arm shoulder extension from 180° and 90° measured on a 1080 Quantum Syncro set to an isokinetic setting for both the concentric and eccentric contraction phases at 30°/second.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron J Mitchell, PhD, Principal Investigator — The University of British Columbia, School of Kinesiology

IPD SHARING:
Plan to Share IPD: No